CLINICAL TRIAL: NCT00926510
Title: Two to Talk: The Use of a Language Toolkit for Toddlers
Brief Title: The Use of a Language Toolkit for Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Michael Steiner, MD, Asst. Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0549
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Language Acquisition

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Language Toolkit (Experimental): Language toolkit composed of simple tools that parents can use to interact with child and help language acquisition.
  Interventions: Behavioral: Language toolkit
- 2 (Placebo Comparator): Safety counseling and smoke detector
  Interventions: Behavioral: Safety counseling

INTERVENTIONS:
Behavioral: Language toolkit — Simple toolkit of interactive things to stimulate language.
  Arms: Language Toolkit
Behavioral: Safety counseling — Smoke detector and general safety counseling
  Arms: 2

SUMMARY:
To investigate whether young children with isolated expressive language delay benefit from early intervention with a simple language toolkit and brief instructions provided to their caregivers.

We hypothesize that children whose families are provided the language toolkit will develop more words over the subsequent 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 14.5 to 18.5 months
* Below average expressive language
* Otherwise normal development

Exclusion Criteria:

* Other developmental delay
* Non-English primary language

Ages: 14 Months to 19 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Language/Words acquisition | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Steiner, MD, Study Director — UNC Hospitals; Jennifer Hartz, MD, Principal Investigator — UNC Hospitals; Mary Ann Cross, MD, Principal Investigator — UNC Hospitals; Karen L Wysocki, MS, M Ed, Study Director — UNC Hospitals
Locations (1):
- North Carolina Children's Hospital, Chapel Hill, North Carolina, United States